CLINICAL TRIAL: NCT01706302
Title: Burden of Respiratory Syncytial Virus (RSV) in the United Kingdom, 1995 to 2009
Brief Title: Burden of Respiratory Syncytial Virus (RSV) in the United Kingdom From 1995 to 2009
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Sage Analytica (Industry)
Responsible Party: Sponsor
Other Study IDs: 116357
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Respiratory Syncyctial Virus Vaccines
Keywords: General Practice Research Database; Burden of Disease; Clinical Practice Research Datalink; Hospital Episode Statistics; Office of National Statistics; RSV
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort Group
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — The previous study has used four primary data sources: the General Practice Research Data (GPRD [recently re-named Clinical Practice Research Datalink (CPRD)], for mild outcomes), the Hospital Episode Statistics database (HES, for hospitalizations), the Office of National Statistics mortality database (ONS, for mortality), and weekly virology data from the Health Protection Agency (HPA). The extracted data are referred to as the EPI-FLU-018 BOD UK DB database. Weekly time series will be generated to estimate the RSV burden and characterize it in terms of incidence of GP consultations, hospitalizations and deaths for each of the respiratory and non-respiratory outcomes (including GP antibiotic prescriptions), stratified by age and risk group.

SUMMARY:
The study will assess the burden of RSV-attributable general practice consultations, hosptializations, and deaths by age and risk group in in United Kingdom from 1995 to 2009.

DETAILED DESCRIPTION:
This epidemiological study is based on an already existing database of time series regression modeling outputs generated during the generated by EPI-FLU-018 BOD UK DB (116273) study, which estimated the burden of influenza in terms of General Practitioner (GP) consultations, hospitalizations, and deaths associated with various respiratory and non-respiratory outcomes.

ELIGIBILITY:
Inclusion Criteria:

• Included in the EPI-FLU-018 BOD UK DB BOD UK DB (eTrack: 116273) study database. The inclusion criterion for EPI-FLU-018 was registration with an acceptable flag in the CPRD, or registration in the HES database or the ONS mortality data with a flu-related event.

Exclusion Criteria:

• Not Applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects included in the 116273 study who were registered with an acceptable flag in the CPRD, or with a potentially RSV-related event in the HES database or the ONS mortality data.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Occurrence in the EPI-FLU-018 BOD UK DB results database of potentially RSV-attributable GP consultation, hospitalization or death associated with respiratory outcomes. | From 1995 to 2009

SECONDARY OUTCOMES:
Occurrence in the EPI-FLU-018 BOD UK DB results database of potentially RSV-attributable GP consultation, hospitalization or death associated with non-respiratory outcomes. | From 1995 to 2009
Occurrence in the EPI-FLU-018 BOD UK DB results database of potentially RSV-attributable GP prescription of antibiotics relevant to respiratory disease, by age and risk group. | From 1995 to 2009
Peak occurrence of potentially RSV-attributable hospitalizations and deaths in elderly and pediatric populations. | From 1995 to 2009
Occurrence of potentially RSV-attributable deaths among the total number of RSV-attributable hospitalizations and cases, by age and risk group. | From 1995 to 2009

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Taylor S, Taylor RJ, Lustig RL, Schuck-Paim C, Haguinet F, Webb DJ, Logie J, Matias G, Fleming DM. Modelling estimates of the burden of respiratory syncytial virus infection in children in the UK. BMJ Open. 2016 Jun 2;6(6):e009337. doi: 10.1136/bmjopen-2015-009337. PMID 27256085
- [Derived] Fleming DM, Taylor RJ, Lustig RL, Schuck-Paim C, Haguinet F, Webb DJ, Logie J, Matias G, Taylor S. Modelling estimates of the burden of Respiratory Syncytial virus infection in adults and the elderly in the United Kingdom. BMC Infect Dis. 2015 Oct 23;15:443. doi: 10.1186/s12879-015-1218-z. PMID 26497750